CLINICAL TRIAL: NCT07402421
Title: Diffusion-Weighted Magnetic Resonance Imaging as a Non-invasive Tool for Differentiating Endometrial Lesions: Accuracy in Comparison With Histopathology
Brief Title: DWI MRI for Differentiating Endometrial Lesions in Comparison With Histopathology
Acronym: MRI in ELs
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nardine Boshra, Resident, Sohag University
Other Study IDs: Soh-Med-26-1-4MS
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Lesions
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected endometrial lesions: This cohort includes women with clinically or radiologically suspected endometrial lesions who undergo pelvic magnetic resonance imaging with diffusion-weighted sequences. Diffusion-weighted MRI findings, including signal characteristics and apparent diffusion coefficient (ADC) values, are evaluated and compared with histopathological examination results obtained from endometrial biopsy or surgical specimens, which serve as the reference standard. No therapeutic intervention is assigned as part of this study.
  Interventions: Other: Diagnostic imaging (DWI MRI) in comparison with histopathology

INTERVENTIONS:
Other: Diagnostic imaging (DWI MRI) in comparison with histopathology — Participants undergo pelvic magnetic resonance imaging including diffusion-weighted imaging sequences as part of routine diagnostic evaluation. Diffusion-weighted MRI is used to assess endometrial lesions by analyzing signal characteristics and apparent diffusion coefficient (ADC) values. No experimental treatment or additional procedures are performed beyond standard clinical care.

SUMMARY:
The aim of this study is to evaluate the diagnostic accuracy of Diffusion Weighted Magnetic Resonance Imaging (DW MRI) in differentiating benign from malignant endometrial lesions, using histopathological examination as the reference standard.

DETAILED DESCRIPTION:
This study is designed to assess the diagnostic performance of diffusion-weighted magnetic resonance imaging (DW-MRI) in the evaluation of endometrial lesions. Women with suspected endometrial pathology who undergo pelvic MRI including diffusion-weighted sequences will be included. DW-MRI findings will be analyzed to characterize endometrial lesions based on signal intensity and apparent diffusion coefficient (ADC) values.

MRI examinations will be performed using standardized imaging protocols. Lesions will be independently assessed by experienced radiologists who are blinded to histopathological results. DW-MRI characteristics suggestive of benign or malignant pathology will be recorded and correlated with final histopathological diagnosis obtained from endometrial biopsy or surgical specimens, which will serve as the reference standard.

Diagnostic accuracy parameters, including sensitivity, specificity, positive predictive value, negative predictive value, and overall accuracy of DW-MRI in differentiating benign from malignant endometrial lesions, will be calculated. ADC values of benign and malignant lesions will be compared to determine optimal cutoff values for malignancy.

The results of this study aim to clarify the role of DW-MRI as a non-invasive imaging tool in the preoperative assessment of endometrial lesions and its potential contribution to improving diagnostic confidence and patient management.

ELIGIBILITY:
Inclusion Criteria:

* Female patients.
* Presenting with abnormal uterine bleeding or suspected endometrial lesions on ultrasound.

Exclusion Criteria:

* Previous treatment (surgery, hormonal therapy, or radiation) for current endometrial pathology.
* Contraindications to MRI (e.g. pacemaker and severe claustrophobia).
* Pregnancy or renal impairment if contrast-enhanced sequences are used.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: This study will include female patients presenting with abnormal uterine bleeding or suspected endometrial lesions detected on transvaginal ultrasound. Eligible participants will undergo pelvic MRI including diffusion-weighted imaging, followed by histopathological confirmation through endometrial biopsy or surgical specimens. Patients with prior treatment for the current endometrial pathology (including surgery, hormonal therapy, or radiotherapy), contraindications to MRI (such as cardiac pacemakers or severe claustrophobia), pregnancy, or renal impairment when contrast-enhanced sequences are required will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Diffusion-Weighted Magnetic Resonance Imaging as a non-invasive tool for differentiating endometrial lesions: Accuracy in comparison with histopathology | From the time of MRI examination until histopathological confirmation following endometrial biopsy or surgery.
  To evaluate the diagnostic accuracy of diffusion-weighted magnetic resonance imaging (DWI-MRI) in differentiating benign from malignant endometrial lesions, using histopathological examination as the reference standard. Accuracy parameters including sensitivity, specificity, positive predictive value, negative predictive value, and overall diagnostic accuracy will be assessed.
Diffusion-Weighted Magnetic Resonance Imaging as a non-invasive tool for differentiating endometrial lesions: Accuracy in comparison with histopathology | From the time of MRI examination until histopathological confirmation following endometrial biopsy or surgery, within a period of up to 4 weeks.
  To evaluate the diagnostic accuracy of diffusion-weighted magnetic resonance imaging (DWI-MRI) in differentiating benign from malignant endometrial lesions, using histopathological examination as the reference standard. Accuracy parameters including sensitivity, specificity, positive predictive value, negative predictive value, and overall diagnostic accuracy will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed T Solyman, MD, Principal Investigator
Locations (1):
- Sohag University Hospital, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy and confidentiality considerations